CLINICAL TRIAL: NCT06898008
Title: Characterization of Children with Complaints of Excessive Daytime Sleepiness
Acronym: CEPSDE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5430
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Excessive Daytime Sleepiness
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — Psychometrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- patient < 18 years of age, having received a diagnostic evaluation for hypersomnia in the HFME sleep
  Interventions: Other: Assessment of socio-demographic, anthropometric, psychometric and clinical characteristics

INTERVENTIONS:
Other: Assessment of socio-demographic, anthropometric, psychometric and clinical characteristics — age, sex and place of residence, socioeconomic level, education, anthropometric data, first-degree family history, screen time, physical activity time, sleep time, comorbidity, drug treatments, education, total IQ, results of Epworth, CDI, ISI, ADHD, CONNERS, SCSC, Horne and Ostberg questionnaires, hearing aids, referring professional, melatonin dosage, ferritinemia, etiology of sleepiness

SUMMARY:
10% of the population suffers from excessive daytime sleepiness. This can be explained by a variety of etiologies: psychiatric disorders, altered sleep quantity or quality, hypersomnia... The consequences on quality of life are not negligible, with emotional, academic, social, financial and somatic repercussions. Diagnosing and managing them is essential. This is the role of the HFME's Child Sleep Service, a reference center for rare narcolepsy and hypersomnia, which carries out a weekly hypersomnia assessment. In this context, the investigators are carrying out a retrospective descriptive study, the primary objective of which is to describe the results and diagnoses of hypersomnia check-ups in the HFME's Sleep Department, in order to obtain feedback on the center's activity and its evolution.

The secondary objectives are to characterize the patients in the different diagnostic groups, to highlight factors associated with the different diagnoses, and to describe changes in patient characteristics over time.

ELIGIBILITY:
Inclusion Criteria:

* - Patient hospitalized in the HFME sleep department for a "diagnostic assessment of hypersomnia".
* Age under 18 at the time of hospitalization
* From January 2015 to December 2023

Exclusion Criteria:

* - No balance sheet
* Age over 18 at time of hospitalization
* Assessment for medicolegal or therapeutic adaptation purposes

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients at the HFME university hospital center, third-line referral center for the Auvergne-Rhônes-Alpes region (France)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Describe the results and diagnoses of hypersomnia assessments in the HFME Sleep Department | Feedback consultation 1 month after inpatient assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'épileptologie clinique, des troubles du sommeil et de neurologie fonctionnelle de l'enfant - Hôpital Femme Mère Enfant, France, Bron, France